CLINICAL TRIAL: NCT01367028
Title: Multicentre Randomized Phase II Study of Neoadjuvant Trastuzumab Plus Docetaxel With and Without Bevacizumab and Trastuzumab Plus Docetaxel Plus Non-pegylated Liposome-encapsulated Doxorubicin (NPLD) With and Without Bevacizumab in HER2-positive Early Breast Cancer
Brief Title: A Phase II Study of Neoadjuvant Trastuzumab+Docetaxel+NPLD+/-Bevacizumab in Her2-pos. Early Breast Cancer
Acronym: ABCSG 32
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Austrian Breast & Colorectal Cancer Study Group (Network)
Collaborators: Hoffmann-La Roche (Industry); Cephalon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABCSG 32; 2010-023324-25 (EudraCT Number)
Record Dates: First submitted 2011-05-31; First posted 2011-06-06 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Breast Cancer
Keywords: HER2-positive early breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Docetaxel; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A: Trastuzumab+Docetaxel (Other)
  Interventions: Drug: Trastuzumab, Docetaxel
- B: Trastuzumab+Docetaxel+Bevacizumab (Experimental)
  Interventions: Drug: Trastuzumab, Docetaxel, Bevacizumab
- C: Trastuzumab+Docetaxel+NPLD (Experimental)
  Interventions: Drug: Trastuzumab+Docetaxel+NPLD
- D: Trastuzumab+Docetaxel+NPLD+Bevacizumab (Experimental)
  Interventions: Drug: Trastuzumab+Docetaxel+NPLD+Bevacizumab

INTERVENTIONS:
Drug: Trastuzumab, Docetaxel — 6 cycles - Day1 (Day22 = Day1): Trastuzumab: 8 mg/kg loading dose (1st cycle) i.v.; 6 mg/kg maintenance dose in subsequent cycles i.v.
  Docetaxel: 100 mg/m2 by 60 min i.v. infusion
  Other Names: Therapy Arm A
  Arms: A: Trastuzumab+Docetaxel
Drug: Trastuzumab, Docetaxel, Bevacizumab — 6 cycles - Day1 (Day22 = Day1): Trastuzumab: 8 mg/kg loading dose (1st cycle) i.v.; 6 mg/kg maintenance dose in subsequent cycles i.v.
  Docetaxel: 100 mg/m2 by 60 min i.v. infusion Bevacizumab 15 mg/kg
  Other Names: Therapy Arm B
  Arms: B: Trastuzumab+Docetaxel+Bevacizumab
Drug: Trastuzumab+Docetaxel+NPLD — 6 cycles - Day1 (Day22=Day1): Trastuzumab: 8 mg/kg loading dose (1st cycle) i.v.; 6 mg/kg maintenance dose in subsequent cycles i.v.
  Docetaxel: 75 mg/m2 by 60 min IV infusion NPLD 50 mg/m2 by 60 min i.v. infusion
  Other Names: Therapy Arm C
  Arms: C: Trastuzumab+Docetaxel+NPLD
Drug: Trastuzumab+Docetaxel+NPLD+Bevacizumab — 6 cycles - Day1 (Day22= Day1): Trastuzumab: 8 mg/kg loading dose (1st cycle) i.v.; 6 mg/kg maintenance dose in subsequent cycles i.v.
  Docetaxel: 75 mg/m2 by 60 min i.v. infusion NPLD: 50 mg/m2 by 60 min i.v. infusion; Bevacizumab 15 mg/kg
  Other Names: Therapy Arm D
  Arms: D: Trastuzumab+Docetaxel+NPLD+Bevacizumab

SUMMARY:
Multicenter randomised phase II study of neoadjuvant therapy in HER2 positive early breast cancer. Primary aim is to evaluate the cardiac toxicity of the combined treatment (trastuzumab, docetaxel, bevacizumab, NPLD) in comparison to the standard therapy.

DETAILED DESCRIPTION:
The target study population consists of male and female pre- and postmenopausal patients with HER2-positive, adenocarcinoma of the breast (except inflammatory breast cancer, T4d) scheduled to receive neoadjuvant cytotoxic treatment.

Patients must have pathologically confirmed breast cancer with histologically confirmed HER2 over-expression. At screening, patients must have an adequate left ventricular ejection fraction (LVEF); an ECOG performance status of 0 or 1; adequate liver, renal and bone marrow function; and be free of other serious diseases that could affect protocol compliance or interpretation of results.

Patients should not be at increased risk of GI perforation, hypertension, proteinuria, wound healing complications, thromboembolism or hemorrhage. Patients must not have had another primary malignancy that could affect compliance with the protocol or interpretation of results. Patients with central nervous system (CNS) metastases are excluded. Pregnant or lactating females are excluded. Patients with hypertension (>150 mmHG systolic or >100 mmHG diastolic) and patients with a history of GI perforation, abdominal fistula or intra-abdominal abscess within 6 months of study entry are excluded.

Full anticoagulation therapy at study entry is allowed as long as the patient has been on a stable level of anticoagulants for at least 2 weeks at the time of study treatment start.

ELIGIBILITY:
Inclusion Criteria:

* Female or male, age ≥ 18 years
* Pathologically confirmed invasive primary breast adenocarcinoma (except inflammatory breast cancer, T4d) scheduled for taxane containing neoadjuvant systemic treatment with/without palpable lymph nodes.
* Documented HER2 protein overexpression as determined by immunohistochemistry (IHC) 3+ or by demonstrated HER2/c-erbB2 gene amplification of the primary tumor by a local laboratory.
* LVEF ≥ 55% measured by echocardiography or MUGA within 4 weeks before randomization
* ECOG Performance Status ≤ 1
* Able and willing to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.
* Written Informed Consent

Exclusion Criteria:

Current Treatment

* Requirement for concurrent use of the antiviral agent sorivudine or chemically related analogues, such as brivudine.
* Chronic daily treatment with corticosteroids excl. inhaled steroids.
* Chronic daily treatment with aspirin and aspirin analogs or clopidogrel
* Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to randomization or anticipation of need for major surgery during the course of study treatment
* Current or recent (within 30 days prior to randomization) treatment with another investigational drug or participation in another investigational study.

Laboratory

* Inadequate bone marrow function
* Inadequate liver function
* Inadequate renal function
* Patients not receiving anticoagulant medication who have activated partial thromboplastin time (aPTT) within 7 days prior to Day1 of the cycle 1.

Concomitant Conditions

* Other malignancy within the last 5 years before randomization except for curatively treated carcinoma in situ of the cervix or non-melanomatous skin cancer
* Evidence of distant metastasis judged clinically and at least by chest-X-ray, liver-sonography and bone scan. If there is any clinical suspicion of brain metastasis, a CT-scan or MRI of the brain must be conducted within 4 weeks prior to randomization.
* Serious concurrent disease which could affect compliance with the protocol or interpretation of results, including, but not limited to:

  * Active infection requiring i.v. antibiotics
  * Uncontrolled hypertension
  * Clinically significant history of cardiovascular disease as indicated by: cerebrovascular accident or stroke; myocardial infarction; unstable angina; NYHA Grade II or greater CHF; cardiac arrhythmia requiring medication; clinically significant valvular heart disease.
  * Dyspnea at rest necessitating supportive oxygen therapy or with significant pleural effusions
  * Poorly controlled diabetes mellitus
  * History or evidence upon physical/neurological examination of CNS disease unrelated to cancer (e.g. uncontrolled seizures) unless adequately treated with standard medical therapy
  * History or evidence of inherited bleeding diathesis or coagulopathy with the risk of bleeding
  * History of abdominal fistula, GI perforation, or intra-abdominal abscess within 6 months of randomization
  * Serious non-healing wound, peptic ulcer, or bone fracture
  * Clinically significant malabsorption syndrome, ulcerative colitis, disease affecting GI function, resection of the stomach or small bowel, or inability to take oral medication
  * Uncorrected hypokalemia or hypomagnesemia
  * Organ allografts requiring immunosuppressive therapy
* Evidence of any other disease, metabolic or psychological dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, may affect patient compliance with study routines, or place the patient at high risk from treatment related complications.
* Known hypersensitivity to any of the study drugs/excipients.
* Hypersensitivity to Chinese hamster ovary cell products or other recombinant human or humanized antibodies.

Other

* Pregnant, lactating females or women of childbearing potential without a negative pregnancy test
* Fertile males or females of childbearing potential
* Patients not accessible for treatment or follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-06; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Cardiac toxicity | between day 1 of cycle 1 and day 28 after the day of final surgery
  to evaluate the cardiac toxicity of the combination trastuzumab+docetaxel+bevacizumab and trastuzumab+docetaxel+NPLD +/- bevacizumab in comparison to the standard therapy, trastuzumab+docetaxel using a composite endpoint appearing between day 1 of cycle 1 and day 28 after the day of final surgery.

SECONDARY OUTCOMES:
Pathological complete response (ypCR) | up to 22 weeks
  ypCR defined as absence of invasive tumor at time of final surgery
Total pathological complete response (ytpCR) | up to 22 weeks
  ytpCR defined as absence of invasive tumor and tumor cells in the breast and the axillar lymphnodes (ypT0 or yDCIS and ypN=0)
Overall clinical response rate (cORR) | up to 22 weeks
  cORR defined as the percentage of patients with either a complete clinical response (cCR) or a partial clinical response (cPR), but no ypCR
Safety evaluation according to patients numbers of AEs, SAEs, lab test abnormalities, cardiac assessment, clinical evaluation | up to 22 weeks
  Safety (AEs, SAEs, lab test abnormalities, cardiac assessment, clinical evaluation)of the combination trastuzumab and docetaxel with bevacizumab and trastuzumab, docetaxel, and NPLD plus/minus bevacizumab at the time of final surgery

CONTACTS AND LOCATIONS:
Overall Officials: Guenther Steger, MD, Principal Investigator — Austrian Breast & Colorectal Cancer Study Group
Locations (11):
- Austria (11):
  - Paracelsus Medical University Salzburg-Oncology, Coop. Group, Salzburg, Salzburg
  - Medical University of Graz-Oncology; Coop. Group, Graz, Styria
  - State Hospital Leoben, Leoben, Styria
  - Gynaegological Medical University Innsbruck, Innsbruck, Tyrol
  - District Hospital Kufstein, Kufstein, Tyrol
  - Hospital BHS Linz, Coop. Study Group, Linz, Upper Austria
  - AKH Linz, Linz, Upper Austria
  - Med. Univ. Vienna; General Hospital Vienna, Vienna, Vienna
  - Medical University Vienna, General Hospital, Vienna, Vienna
  - State Hospital Vienna-Hietzing, Vienna, Vienna
  - State Hospital Feldkirch, Coop. Group, Feldkirch, Vorarlberg

REFERENCES:
- [Background] Chan S, Davidson N, Juozaityte E, Erdkamp F, Pluzanska A, Azarnia N, Lee LW. Phase III trial of liposomal doxorubicin and cyclophosphamide compared with epirubicin and cyclophosphamide as first-line therapy for metastatic breast cancer. Ann Oncol. 2004 Oct;15(10):1527-34. doi: 10.1093/annonc/mdh393. PMID 15367414
- [Background] Clark GM, Sledge GW Jr, Osborne CK, McGuire WL. Survival from first recurrence: relative importance of prognostic factors in 1,015 breast cancer patients. J Clin Oncol. 1987 Jan;5(1):55-61. doi: 10.1200/JCO.1987.5.1.55. PMID 3806159
- [Background] Cobleigh MA, Langmuir VK, Sledge GW, Miller KD, Haney L, Novotny WF, Reimann JD, Vassel A. A phase I/II dose-escalation trial of bevacizumab in previously treated metastatic breast cancer. Semin Oncol. 2003 Oct;30(5 Suppl 16):117-24. doi: 10.1053/j.seminoncol.2003.08.013. PMID 14613032
- [Background] Coleman MP, Gatta G, Verdecchia A, Esteve J, Sant M, Storm H, Allemani C, Ciccolallo L, Santaquilani M, Berrino F; EUROCARE Working Group. EUROCARE-3 summary: cancer survival in Europe at the end of the 20th century. Ann Oncol. 2003;14 Suppl 5:v128-49. doi: 10.1093/annonc/mdg756. No abstract available. PMID 14684503
- [Background] Cortes J, Di Cosimo S, Climent MA, Cortes-Funes H, Lluch A, Gascon P, Mayordomo JI, Gil M, Benavides M, Cirera L, Ojeda B, Rodriguez CA, Trigo JM, Vazquez J, Regueiro P, Dorado JF, Baselga J; Spanish Breast Cancer Cooperative Group SOLTI. Nonpegylated liposomal doxorubicin (TLC-D99), paclitaxel, and trastuzumab in HER-2-overexpressing breast cancer: a multicenter phase I/II study. Clin Cancer Res. 2009 Jan 1;15(1):307-14. doi: 10.1158/1078-0432.CCR-08-1113. PMID 19118059
- [Background] Crown J, O'Leary M, Ooi WS. Docetaxel and paclitaxel in the treatment of breast cancer: a review of clinical experience. Oncologist. 2004;9 Suppl 2:24-32. doi: 10.1634/theoncologist.9-suppl_2-24. PMID 15161988
- [Background] Eskens FA. Angiogenesis inhibitors in clinical development; where are we now and where are we going? Br J Cancer. 2004 Jan 12;90(1):1-7. doi: 10.1038/sj.bjc.6601401. PMID 14710197
- [Background] Ferrara N, Davis-Smyth T. The biology of vascular endothelial growth factor. Endocr Rev. 1997 Feb;18(1):4-25. doi: 10.1210/edrv.18.1.0287. No abstract available. PMID 9034784
- [Background] Ferrara N, Henzel WJ. Pituitary follicular cells secrete a novel heparin-binding growth factor specific for vascular endothelial cells. Biochem Biophys Res Commun. 1989 Jun 15;161(2):851-8. doi: 10.1016/0006-291x(89)92678-8. PMID 2735925
- [Background] Ferrara N. Vascular endothelial growth factor as a target for anticancer therapy. Oncologist. 2004;9 Suppl 1:2-10. doi: 10.1634/theoncologist.9-suppl_1-2. PMID 15178810
- [Background] Folkman J. What is the role of thymidine phosphorylase in tumor angiogenesis. J Natl Cancer Inst. 1996 Aug 21;88(16):1091-2. doi: 10.1093/jnci/88.16.1091. No abstract available. PMID 8757181
- [Background] Fountzilas G, Razis E, Tsavdaridis D, Karina M, Labropoulos S, Christodoulou C, Mavroudis D, Gogas H, Georgoulias V, Skarlos D. Continuation of trastuzumab beyond disease progression is feasible and safe in patients with metastatic breast cancer: a retrospective analysis of 80 cases by the hellenic cooperative oncology group. Clin Breast Cancer. 2003 Jun;4(2):120-5. doi: 10.3816/cbc.2003.n.017. PMID 12864940
- [Background] Gelmon KA, Mackey J, Verma S, Gertler SZ, Bangemann N, Klimo P, Schneeweiss A, Bremer K, Soulieres D, Tonkin K, Bell R, Heinrich B, Grenier D, Dias R. Use of trastuzumab beyond disease progression: observations from a retrospective review of case histories. Clin Breast Cancer. 2004 Apr;5(1):52-8; discussion 59-62. doi: 10.3816/cbc.2004.n.010. PMID 15140285
- [Background] Gerber HP, Ferrara N. Pharmacology and pharmacodynamics of bevacizumab as monotherapy or in combination with cytotoxic therapy in preclinical studies. Cancer Res. 2005 Feb 1;65(3):671-80. PMID 15705858
- [Background] Giordano SH, Duan Z, Kuo YF, Hortobagyi GN, Freeman J, Goodwin JS. Impact of a scientific presentation on community treatment patterns for primary breast cancer. J Natl Cancer Inst. 2006 Mar 15;98(6):382-8. doi: 10.1093/jnci/djj090. PMID 16537830
- [Background] Greene FL, Page DL Fleming ID et al. eds. AJCC Cancer Staging Handbook. 6th Edition. 2002; Springer
- [Background] Griffiths L, Dachs GU, Bicknell R, Harris AL, Stratford IJ. The influence of oxygen tension and pH on the expression of platelet-derived endothelial cell growth factor/thymidine phosphorylase in human breast tumor cells grown in vitro and in vivo. Cancer Res. 1997 Feb 15;57(4):570-2. PMID 9044826
- [Background] Harris L, Batist G, Belt R, Rovira D, Navari R, Azarnia N, Welles L, Winer E; TLC D-99 Study Group. Liposome-encapsulated doxorubicin compared with conventional doxorubicin in a randomized multicenter trial as first-line therapy of metastatic breast carcinoma. Cancer. 2002 Jan 1;94(1):25-36. doi: 10.1002/cncr.10201. PMID 11815957
- [Background] Hicklin DJ, Ellis LM. Role of the vascular endothelial growth factor pathway in tumor growth and angiogenesis. J Clin Oncol. 2005 Feb 10;23(5):1011-27. doi: 10.1200/JCO.2005.06.081. Epub 2004 Dec 7. PMID 15585754
- [Background] Bonneterre ME, Bonneterre J. Reply to the article
- [Background] Hirsh J, Raschke R. Heparin and low-molecular-weight heparin: the Seventh ACCP Conference on Antithrombotic and Thrombolytic Therapy. Chest. 2004 Sep;126(3 Suppl):188S-203S. doi: 10.1378/chest.126.3_suppl.188S. PMID 15383472
- [Background] Hotchkiss KA, Ashton AW, Mahmood R, Russell RG, Sparano JA, Schwartz EL. Inhibition of endothelial cell function in vitro and angiogenesis in vivo by docetaxel (Taxotere): association with impaired repositioning of the microtubule organizing center. Mol Cancer Ther. 2002 Nov;1(13):1191-200. PMID 12479700
- [Background] Itakura J, Ishiwata T, Shen B, Kornmann M, Korc M. Concomitant over-expression of vascular endothelial growth factor and its receptors in pancreatic cancer. Int J Cancer. 2000 Jan 1;85(1):27-34. doi: 10.1002/(sici)1097-0215(20000101)85:13.0.co;2-8. PMID 10585578
- [Background] Izumi Y, Xu L, di Tomaso E, Fukumura D, Jain RK. Tumour biology: herceptin acts as an anti-angiogenic cocktail. Nature. 2002 Mar 21;416(6878):279-80. doi: 10.1038/416279b. PMID 11907566
- [Background] Jain D. Cardiotoxicity of doxorubicin and other anthracycline derivatives. J Nucl Cardiol. 2000 Jan-Feb;7(1):53-62. doi: 10.1067/mnc.2000.103324. No abstract available. PMID 10698235
- [Background] Jain RK. Normalizing tumor vasculature with anti-angiogenic therapy: a new paradigm for combination therapy. Nat Med. 2001 Sep;7(9):987-9. doi: 10.1038/nm0901-987. No abstract available. PMID 11533692
- [Background] Jiang BH, Agani F, Passaniti A, Semenza GL. V-SRC induces expression of hypoxia-inducible factor 1 (HIF-1) and transcription of genes encoding vascular endothelial growth factor and enolase 1: involvement of HIF-1 in tumor progression. Cancer Res. 1997 Dec 1;57(23):5328-35. PMID 9393757
- [Background] Jones SE, Erban J, Overmoyer B, Budd GT, Hutchins L, Lower E, Laufman L, Sundaram S, Urba WJ, Pritchard KI, Mennel R, Richards D, Olsen S, Meyers ML, Ravdin PM. Randomized phase III study of docetaxel compared with paclitaxel in metastatic breast cancer. J Clin Oncol. 2005 Aug 20;23(24):5542-51. doi: 10.1200/JCO.2005.02.027. PMID 16110015
- [Background] Kerbel RS, Kamen BA. The anti-angiogenic basis of metronomic chemotherapy. Nat Rev Cancer. 2004 Jun;4(6):423-36. doi: 10.1038/nrc1369. No abstract available. PMID 15170445
- [Background] Kieser A, Weich HA, Brandner G, Marme D, Kolch W. Mutant p53 potentiates protein kinase C induction of vascular endothelial growth factor expression. Oncogene. 1994 Mar;9(3):963-9. PMID 8108142
- [Background] Kim KJ, Li B, Winer J, Armanini M, Gillett N, Phillips HS, Ferrara N. Inhibition of vascular endothelial growth factor-induced angiogenesis suppresses tumour growth in vivo. Nature. 1993 Apr 29;362(6423):841-4. doi: 10.1038/362841a0. PMID 7683111
- [Background] Klement G, Baruchel S, Rak J, Man S, Clark K, Hicklin DJ, Bohlen P, Kerbel RS. Continuous low-dose therapy with vinblastine and VEGF receptor-2 antibody induces sustained tumor regression without overt toxicity. J Clin Invest. 2000 Apr;105(8):R15-24. doi: 10.1172/JCI8829. PMID 10772661
- [Background] Konecny GE, Meng YG, Untch M, Wang HJ, Bauerfeind I, Epstein M, Stieber P, Vernes JM, Gutierrez J, Hong K, Beryt M, Hepp H, Slamon DJ, Pegram MD. Association between HER-2/neu and vascular endothelial growth factor expression predicts clinical outcome in primary breast cancer patients. Clin Cancer Res. 2004 Mar 1;10(5):1706-16. doi: 10.1158/1078-0432.ccr-0951-3. PMID 15014023
- [Background] Lee CG, Heijn M, di Tomaso E, Griffon-Etienne G, Ancukiewicz M, Koike C, Park KR, Ferrara N, Jain RK, Suit HD, Boucher Y. Anti-Vascular endothelial growth factor treatment augments tumor radiation response under normoxic or hypoxic conditions. Cancer Res. 2000 Oct 1;60(19):5565-70. PMID 11034104
- [Background] Leyland-Jones B, Gelmon K, Ayoub JP, Arnold A, Verma S, Dias R, Ghahramani P. Pharmacokinetics, safety, and efficacy of trastuzumab administered every three weeks in combination with paclitaxel. J Clin Oncol. 2003 Nov 1;21(21):3965-71. doi: 10.1200/JCO.2003.12.109. Epub 2003 Sep 24. PMID 14507946
- [Background] Linderholm BK, Lindahl T, Holmberg L, Klaar S, Lennerstrand J, Henriksson R, Bergh J. The expression of vascular endothelial growth factor correlates with mutant p53 and poor prognosis in human breast cancer. Cancer Res. 2001 Mar 1;61(5):2256-60. PMID 11280795
- [Background] Liu CD, Tilch L, Kwan D, McFadden DW. Vascular endothelial growth factor is increased in ascites from metastatic pancreatic cancer. J Surg Res. 2002 Jan;102(1):31-4. doi: 10.1006/jsre.2001.6307. PMID 11792148
- [Background] Marty M, Espie M, Cottu PH, Cuvier C, Lerebours F. Optimizing chemotherapy for patients with advanced breast cancer. Oncology. 1999 Jul;57 Suppl 1:21-6. doi: 10.1159/000055265. PMID 10436413
- [Background] Marty M, Cognetti F, Maraninchi D, Snyder R, Mauriac L, Tubiana-Hulin M, Chan S, Grimes D, Anton A, Lluch A, Kennedy J, O'Byrne K, Conte P, Green M, Ward C, Mayne K, Extra JM. Randomized phase II trial of the efficacy and safety of trastuzumab combined with docetaxel in patients with human epidermal growth factor receptor 2-positive metastatic breast cancer administered as first-line treatment: the M77001 study group. J Clin Oncol. 2005 Jul 1;23(19):4265-74. doi: 10.1200/JCO.2005.04.173. Epub 2005 May 23. PMID 15911866
- [Background] Mayer LD, Tai LC, Ko DS, Masin D, Ginsberg RS, Cullis PR, Bally MB. Influence of vesicle size, lipid composition, and drug-to-lipid ratio on the biological activity of liposomal doxorubicin in mice. Cancer Res. 1989 Nov 1;49(21):5922-30. PMID 2790807
- [Background] Menard S, Casalini P, Tomasic G, Pilotti S, Cascinelli N, Bufalino R, Perrone F, Longhi C, Rilke F, Colnaghi MI. Pathobiologic identification of two distinct breast carcinoma subsets with diverging clinical behaviors. Breast Cancer Res Treat. 1999 May;55(2):169-77. doi: 10.1023/a:1006262324959. PMID 10481944
- [Background] Miller KD, Chap LI, Holmes FA, Cobleigh MA, Marcom PK, Fehrenbacher L, Dickler M, Overmoyer BA, Reimann JD, Sing AP, Langmuir V, Rugo HS. Randomized phase III trial of capecitabine compared with bevacizumab plus capecitabine in patients with previously treated metastatic breast cancer. J Clin Oncol. 2005 Feb 1;23(4):792-9. doi: 10.1200/JCO.2005.05.098. PMID 15681523
- [Background] Miller K, Wang M, Gralow J, Dickler M, Cobleigh M, Perez EA, Shenkier T, Cella D, Davidson NE. Paclitaxel plus bevacizumab versus paclitaxel alone for metastatic breast cancer. N Engl J Med. 2007 Dec 27;357(26):2666-76. doi: 10.1056/NEJMoa072113. PMID 18160686
- [Background] Miwa M, Ura M, Nishida M, Sawada N, Ishikawa T, Mori K, Shimma N, Umeda I, Ishitsuka H. Design of a novel oral fluoropyrimidine carbamate, capecitabine, which generates 5-fluorouracil selectively in tumours by enzymes concentrated in human liver and cancer tissue. Eur J Cancer. 1998 Jul;34(8):1274-81. doi: 10.1016/s0959-8049(98)00058-6. PMID 9849491
- [Background] Moghaddam A, Zhang HT, Fan TP, Hu DE, Lees VC, Turley H, Fox SB, Gatter KC, Harris AL, Bicknell R. Thymidine phosphorylase is angiogenic and promotes tumor growth. Proc Natl Acad Sci U S A. 1995 Feb 14;92(4):998-1002. doi: 10.1073/pnas.92.4.998. PMID 7532308
- [Background] Mross K, Niemann B, Massing U, Drevs J, Unger C, Bhamra R, Swenson CE. Pharmacokinetics of liposomal doxorubicin (TLC-D99; Myocet) in patients with solid tumors: an open-label, single-dose study. Cancer Chemother Pharmacol. 2004 Dec;54(6):514-24. doi: 10.1007/s00280-004-0825-y. Epub 2004 Aug 21. PMID 15322827
- [Background] Mukhopadhyay D, Tsiokas L, Sukhatme VP. Wild-type p53 and v-Src exert opposing influences on human vascular endothelial growth factor gene expression. Cancer Res. 1995 Dec 15;55(24):6161-5. PMID 8521408
- [Background] Paterson MC, Dietrich KD, Danyluk J, Paterson AH, Lees AW, Jamil N, Hanson J, Jenkins H, Krause BE, McBlain WA, et al. Correlation between c-erbB-2 amplification and risk of recurrent disease in node-negative breast cancer. Cancer Res. 1991 Jan 15;51(2):556-67. PMID 1670762
- [Background] Petit AM, Rak J, Hung MC, Rockwell P, Goldstein N, Fendly B, Kerbel RS. Neutralizing antibodies against epidermal growth factor and ErbB-2/neu receptor tyrosine kinases down-regulate vascular endothelial growth factor production by tumor cells in vitro and in vivo: angiogenic implications for signal transduction therapy of solid tumors. Am J Pathol. 1997 Dec;151(6):1523-30. PMID 9403702
- [Background] Piccart M. Treatment of advanced breast cancer: current status. Anticancer Drugs. 1996 Aug;7 Suppl 2:5-7. PMID 8862702
- [Background] Piccart MJ, Di Leo A. Future perspectives of docetaxel (Taxotere) in front-line therapy. Semin Oncol. 1997 Aug;24(4 Suppl 10):S10-27-S10-33. PMID 9275004
- [Background] Rak J, Mitsuhashi Y, Bayko L, Filmus J, Shirasawa S, Sasazuki T, Kerbel RS. Mutant ras oncogenes upregulate VEGF/VPF expression: implications for induction and inhibition of tumor angiogenesis. Cancer Res. 1995 Oct 15;55(20):4575-80. PMID 7553632
- [Background] Ramaswamy B, Elias AD, Kelbick NT, Dodley A, Morrow M, Hauger M, Allen J, Rhoades C, Kendra K, Chen HX, Eckhardt SG, Shapiro CL. Phase II trial of bevacizumab in combination with weekly docetaxel in metastatic breast cancer patients. Clin Cancer Res. 2006 May 15;12(10):3124-9. doi: 10.1158/1078-0432.CCR-05-2603. PMID 16707611
- [Background] Relf M, LeJeune S, Scott PA, Fox S, Smith K, Leek R, Moghaddam A, Whitehouse R, Bicknell R, Harris AL. Expression of the angiogenic factors vascular endothelial cell growth factor, acidic and basic fibroblast growth factor, tumor growth factor beta-1, platelet-derived endothelial cell growth factor, placenta growth factor, and pleiotrophin in human primary breast cancer and its relation to angiogenesis. Cancer Res. 1997 Mar 1;57(5):963-9. PMID 9041202
- [Background] Romond EH, Perez EA, Bryant J, Suman VJ, Geyer CE Jr, Davidson NE, Tan-Chiu E, Martino S, Paik S, Kaufman PA, Swain SM, Pisansky TM, Fehrenbacher L, Kutteh LA, Vogel VG, Visscher DW, Yothers G, Jenkins RB, Brown AM, Dakhil SR, Mamounas EP, Lingle WL, Klein PM, Ingle JN, Wolmark N. Trastuzumab plus adjuvant chemotherapy for operable HER2-positive breast cancer. N Engl J Med. 2005 Oct 20;353(16):1673-84. doi: 10.1056/NEJMoa052122. PMID 16236738
- [Background] Ross JS, Fletcher JA. The HER-2/neu oncogene in breast cancer: prognostic factor, predictive factor, and target for therapy. Stem Cells. 1998;16(6):413-28. doi: 10.1002/stem.160413. PMID 9831867
- [Background] Schaller G, Fuchs I, Gonsch T, Weber J, Kleine-Tebbe A, Klare P, Hindenburg HJ, Lakner V, Hinke A, Bangemann N. Phase II study of capecitabine plus trastuzumab in human epidermal growth factor receptor 2 overexpressing metastatic breast cancer pretreated with anthracyclines or taxanes. J Clin Oncol. 2007 Aug 1;25(22):3246-50. doi: 10.1200/JCO.2006.09.6826. Epub 2007 Jun 18. PMID 17577021
- [Background] Shaked Y, Bertolini F, Man S, Rogers MS, Cervi D, Foutz T, Rawn K, Voskas D, Dumont DJ, Ben-David Y, Lawler J, Henkin J, Huber J, Hicklin DJ, D'Amato RJ, Kerbel RS. Genetic heterogeneity of the vasculogenic phenotype parallels angiogenesis; Implications for cellular surrogate marker analysis of antiangiogenesis. Cancer Cell. 2005 Jan;7(1):101-11. doi: 10.1016/j.ccr.2004.11.023. PMID 15652753
- [Background] Sliwkowski MX, Lofgren JA, Lewis GD, Hotaling TE, Fendly BM, Fox JA. Nonclinical studies addressing the mechanism of action of trastuzumab (Herceptin). Semin Oncol. 1999 Aug;26(4 Suppl 12):60-70. PMID 10482195
- [Background] Stemmler HJ, Kahlert S, Siekiera W, Untch M, Heinrich B, Heinemann V. Prolonged survival of patients receiving trastuzumab beyond disease progression for HER2 overexpressing metastatic breast cancer (MBC). Onkologie. 2005 Nov;28(11):582-6. doi: 10.1159/000088296. PMID 16249644
- [Background] Sumizawa T, Furukawa T, Haraguchi M, Yoshimura A, Takeyasu A, Ishizawa M, Yamada Y, Akiyama S. Thymidine phosphorylase activity associated with platelet-derived endothelial cell growth factor. J Biochem. 1993 Jul;114(1):9-14. doi: 10.1093/oxfordjournals.jbchem.a124146. PMID 8407883
- [Background] Sweeney CJ, Miller KD, Sissons SE, Nozaki S, Heilman DK, Shen J, Sledge GW Jr. The antiangiogenic property of docetaxel is synergistic with a recombinant humanized monoclonal antibody against vascular endothelial growth factor or 2-methoxyestradiol but antagonized by endothelial growth factors. Cancer Res. 2001 Apr 15;61(8):3369-72. PMID 11309294
- [Background] Swenson CE, Bolcsak LE, Batist G, Guthrie TH Jr, Tkaczuk KH, Boxenbaum H, Welles L, Chow SC, Bhamra R, Chaikin P. Pharmacokinetics of doxorubicin administered i.v. as Myocet (TLC D-99; liposome-encapsulated doxorubicin citrate) compared with conventional doxorubicin when given in combination with cyclophosphamide in patients with metastatic breast cancer. Anticancer Drugs. 2003 Mar;14(3):239-46. doi: 10.1097/00001813-200303000-00008. PMID 12634619
- [Background] Theodoulou M, Batist G, Campos S, Winer E, Welles L, Hudis C. Phase I study of nonpegylated liposomal doxorubicin plus trastuzumab in patients with HER2-positive breast cancer. Clin Breast Cancer. 2009 May;9(2):101-7. doi: 10.3816/CBC.2009.n.019. PMID 19433391
- [Background] Toi M, Hoshina S, Taniguchi T, Yamamoto Y, Ishitsuka H, Tominaga T. Expression of platelet-derived endothelial cell growth factor/thymidine phosphorylase in human breast cancer. Int J Cancer. 1995 Apr 21;64(2):79-82. doi: 10.1002/ijc.2910640202. PMID 7542228
- [Background] Tong RT, Boucher Y, Kozin SV, Winkler F, Hicklin DJ, Jain RK. Vascular normalization by vascular endothelial growth factor receptor 2 blockade induces a pressure gradient across the vasculature and improves drug penetration in tumors. Cancer Res. 2004 Jun 1;64(11):3731-6. doi: 10.1158/0008-5472.CAN-04-0074. PMID 15172975
- [Background] Tripathy D, Slamon DJ, Cobleigh M, Arnold A, Saleh M, Mortimer JE, Murphy M, Stewart SJ. Safety of treatment of metastatic breast cancer with trastuzumab beyond disease progression. J Clin Oncol. 2004 Mar 15;22(6):1063-70. doi: 10.1200/JCO.2004.06.557. PMID 15020607
- [Background] Vukelja SJ, Lombardo FA, James WD, Weiss RB. Pyridoxine for the palmar-plantar erythrodysesthesia syndrome. Ann Intern Med. 1989 Oct 15;111(8):688-9. doi: 10.7326/0003-4819-111-8-688. No abstract available. PMID 2529807
- [Background] Vukelja SJ, Baker WJ, Burris HA 3rd, Keeling JH, Von Hoff D. Pyridoxine therapy for palmar-plantar erythrodysesthesia associated with taxotere. J Natl Cancer Inst. 1993 Sep 1;85(17):1432-3. doi: 10.1093/jnci/85.17.1432. No abstract available. PMID 8102408
- [Background] Warren RS, Yuan H, Matli MR, Gillett NA, Ferrara N. Regulation by vascular endothelial growth factor of human colon cancer tumorigenesis in a mouse model of experimental liver metastasis. J Clin Invest. 1995 Apr;95(4):1789-97. doi: 10.1172/JCI117857. PMID 7535799
- [Background] Xeloda® (Capecitabine) Investigator Brochure, 9th Version August 2007
- [Background] Yap R, Veliceasa D, Emmenegger U, Kerbel RS, McKay LM, Henkin J, Volpert OV. Metronomic low-dose chemotherapy boosts CD95-dependent antiangiogenic effect of the thrombospondin peptide ABT-510: a complementation antiangiogenic strategy. Clin Cancer Res. 2005 Sep 15;11(18):6678-85. doi: 10.1158/1078-0432.CCR-05-0621. PMID 16166447
- [Background] Yen L, You XL, Al Moustafa AE, Batist G, Hynes NE, Mader S, Meloche S, Alaoui-Jamali MA. Heregulin selectively upregulates vascular endothelial growth factor secretion in cancer cells and stimulates angiogenesis. Oncogene. 2000 Jul 20;19(31):3460-9. doi: 10.1038/sj.onc.1203685. PMID 10918604
- [Result] Amadori D, Gasparini G, Ardizzoni A, Comella G, Saracchini S, Barone C, Bordonaro R, et al. Phase II study of liposomal doxorubicin (Myocet®), docetaxel and trastuzumab combination as first line treatment of patients with HER-2/neu positive locally advanced or metastatic breast cancer. Cancer Res 2009; 69 (Suppl.): (2).January 15, 3149
- [Result] Ansell J, Hirsh J, Poller L, Bussey H, Jacobson A, Hylek E. The pharmacology and management of the vitamin K antagonists: the Seventh ACCP Conference on Antithrombotic and Thrombolytic Therapy. Chest. 2004 Sep;126(3 Suppl):204S-233S. doi: 10.1378/chest.126.3_suppl.204S. PMID 15383473
- [Result] Antón A, Ruiz-Simón A, Plazaola A, Calvo L, Segui M. A, Santabella A, Muňoz M, et al. Phase II study of a 3-weekly liposome-encapsulated doxorubicin/docetaxel/pegfilgrastim in combination with weekly trastuzumab as primary treatment in HER2 positive (HER+) early stage cancer patients (II-IIIa). GEICAM 2003-03 study. Cancer Res 2009; 69 (Suppl.): (2).January 15, 5117
- [Result] Avastin® (Bevacizumab) Investigator Brochure, Fifteenth Version: November 2007
- [Result] Balazsovits JA, Mayer LD, Bally MB, Cullis PR, McDonell M, Ginsberg RS, Falk RE. Analysis of the effect of liposome encapsulation on the vesicant properties, acute and cardiac toxicities, and antitumor efficacy of doxorubicin. Cancer Chemother Pharmacol. 1989;23(2):81-6. doi: 10.1007/BF00273522. PMID 2491964
- [Result] Bartsch R, Wenzel C, Hussian D, Pluschnig U, Sevelda U, Koestler W, Altorjai G, Locker GJ, Mader R, Zielinski CC, Steger GG. Analysis of trastuzumab and chemotherapy in advanced breast cancer after the failure of at least one earlier combination: an observational study. BMC Cancer. 2006 Mar 15;6:63. doi: 10.1186/1471-2407-6-63. PMID 16539726
- [Result] Bartsch R, Wenzel C, Altorjai G, Pluschnig U, Rudas M, Mader RM, Gnant M, Zielinski CC, Steger GG. Capecitabine and trastuzumab in heavily pretreated metastatic breast cancer. J Clin Oncol. 2007 Sep 1;25(25):3853-8. doi: 10.1200/JCO.2007.11.9776. Epub 2007 Aug 6. PMID 17679724
- [Result] Barton GJ, Ponting CP, Spraggon G, Finnis C, Sleep D. Human platelet-derived endothelial cell growth factor is homologous to Escherichia coli thymidine phosphorylase. Protein Sci. 1992 May;1(5):688-90. doi: 10.1002/pro.5560010514. No abstract available. PMID 1304367
- [Result] Batist G, Ramakrishnan G, Rao CS, Chandrasekharan A, Gutheil J, Guthrie T, Shah P, Khojasteh A, Nair MK, Hoelzer K, Tkaczuk K, Park YC, Lee LW. Reduced cardiotoxicity and preserved antitumor efficacy of liposome-encapsulated doxorubicin and cyclophosphamide compared with conventional doxorubicin and cyclophosphamide in a randomized, multicenter trial of metastatic breast cancer. J Clin Oncol. 2001 Mar 1;19(5):1444-54. doi: 10.1200/JCO.2001.19.5.1444. PMID 11230490
- [Result] Bertolini F, Paul S, Mancuso P, Monestiroli S, Gobbi A, Shaked Y, Kerbel RS. Maximum tolerable dose and low-dose metronomic chemotherapy have opposite effects on the mobilization and viability of circulating endothelial progenitor cells. Cancer Res. 2003 Aug 1;63(15):4342-6. PMID 12907602
- [Result] Blum JL, Dieras V, Lo Russo PM, Horton J, Rutman O, Buzdar A, Osterwalder B. Multicenter, Phase II study of capecitabine in taxane-pretreated metastatic breast carcinoma patients. Cancer. 2001 Oct 1;92(7):1759-68. doi: 10.1002/1097-0142(20011001)92:73.0.co;2-a. PMID 11745247
- [Result] Blum JL, Jones SE, Buzdar AU, LoRusso PM, Kuter I, Vogel C, Osterwalder B, Burger HU, Brown CS, Griffin T. Multicenter phase II study of capecitabine in paclitaxel-refractory metastatic breast cancer. J Clin Oncol. 1999 Feb;17(2):485-93. doi: 10.1200/JCO.1999.17.2.485. PMID 10080589
- [Result] Borgstrom P, Gold DP, Hillan KJ, Ferrara N. Importance of VEGF for breast cancer angiogenesis in vivo: implications from intravital microscopy of combination treatments with an anti-VEGF neutralizing monoclonal antibody and doxorubicin. Anticancer Res. 1999 Sep-Oct;19(5B):4203-14. PMID 10628376
- [Result] Budman DR, Meropol NJ, Reigner B, Creaven PJ, Lichtman SM, Berghorn E, Behr J, Gordon RJ, Osterwalder B, Griffin T. Preliminary studies of a novel oral fluoropyrimidine carbamate: capecitabine. J Clin Oncol. 1998 May;16(5):1795-802. doi: 10.1200/JCO.1998.16.5.1795. PMID 9586893
- [Result] Phase II trial of the anti-VEGF antibody bevacizumab in combination with vinorelbine for refractory advanced breast cancer [abstract 446]. Breast Cancer Res Treat 2002;76:S115
- [Result] Browder T, Butterfield CE, Kraling BM, Shi B, Marshall B, O'Reilly MS, Folkman J. Antiangiogenic scheduling of chemotherapy improves efficacy against experimental drug-resistant cancer. Cancer Res. 2000 Apr 1;60(7):1878-86. PMID 10766175
- [Result] Chan S, Friedrichs K, Noel D, Pinter T, Van Belle S, Vorobiof D, Duarte R, Gil Gil M, Bodrogi I, Murray E, Yelle L, von Minckwitz G, Korec S, Simmonds P, Buzzi F, Gonzalez Mancha R, Richardson G, Walpole E, Ronzoni M, Murawsky M, Alakl M, Riva A, Crown J; 303 Study Group. Prospective randomized trial of docetaxel versus doxorubicin in patients with metastatic breast cancer. J Clin Oncol. 1999 Aug;17(8):2341-54. doi: 10.1200/JCO.1999.17.8.2341. PMID 10561296
- [Result] Epstein M, Ayala R, Tchekmedyian N et al. HER-2/neu-overexpressing human breast cancer xenografts exhibit increased angiogenic potential mediated by vascular endothelial growth factor (VEGF). Breast Cancer Res. Treat. 2002; 76: S143
- [Result] Extra JM, Antoine EC, Vincent-Salomon A et al. Favourable effect of trastuzumab (Herceptin®) treatment in metastatic breast cancer patients: results from the French Hermine cohort study. Poster presentation, 2006 SABCS, San Antonio, Texas
- [Result] Hambleton J, Novotny F, Hurwitz H et al. Bevacizumab (Avastin) does not increase the incidence of bleeding in patients with metastatic colorectal cancer receiving simultaneous anticoagulation. ASCO New Orleans 2004,Abstract 3528
- [Result] Herceptin® (Trastuzumab) Investigator Brochure, Version: October 5, 2007
- [Result] Jackisch C, Eustermann H, Schoenegg W et al. Routine clinical usage of trastuzumab (Herceptin®) in advanced breast cancer in Germany from 2001 to 2006. 2007; Poster Presentation, SABCS
- [Result] Jain RK. Antiangiogenic therapy for cancer: current and emerging concepts. Oncology (Williston Park). 2005 Apr;19(4 Suppl 3):7-16. PMID 15934498
- [Result] Kabbinavar FF, Wong JT, Ayala RE et al. The effect of antibody to vascular endothelia growth factor and cisplatin on the growth of lung tumors in nude mice [abstract]. Proc Am Assoc Cancer Res 1995; 36:488
- [Result] Ménard S (on behalf of the Demetra Group). Observational Demetra study: Survival of metastatic breast carcinoma patients after treatment with trastuzumab. J Clin Oncol 26: 2008 (May 20 suppl; abstr 1062)
- [Result] Miles D, Chan A, Romieu G et al. Randomized, double-blind, placebo-controlled, phase III study of bevacizumab with docetaxel or docetaxel with placebo as first-line therapy for patients with locally recurrent or metastatic breast cancer (mBC): AVADO. J Clin Oncol 26:2008 (May 20 Suppl; abstr LBA1011). Presented at the 2008 ASCO Annual Meeting
- [Result] Myers CE. Anthracyclines. In: Chabner B, ed. Pharmacologic principles of cancer treatment. Philadelphia: Saunders 1982: xii, 457 p
- [Result] O'Shaughnessy J, Blackwell KL, Burstein H et al. A randomized study of lapatinib alone or in combination with trastuzumab in heavily pretreated HER2+ metastatic breast cancer progressing on trastuzumab therapy. J Clin Oncol 26: 2008 (May 20 suppl; abstr 1015)
- [Result] Pegram MD, Reese DM. Combined biological therapy of breast cancer using monoclonal antibodies directed against HER2/neu protein and vascular endothelial growth factor. Semin Oncol. 2002 Jun;29(3 Suppl 11):29-37. doi: 10.1053/sonc.2002.34053. PMID 12138395
- [Result] Pegram M, Chan D, Dichmann RA et al., Phase II combined biological therapy targeting the HER2 proto-oncogene and the vascular endothelial growth factor using trastuzumab (T) and bevacizumab (B) as first-line treatment of HER2-amplified breast cancer. 2006; Poster Presentation, SABCS
- [Result] Potchoiba MJ, West M, Smolarek TA, Macaione G, Santacroce E, Lundeen GR. Tissue distribution of doxorubicin in the free and liposomal forms in male Beagles. Proc Am Assoc Cancer Res 1996; 37:A2675
- [Result] Rugo H, Dickler MN, Scott JH et al. Change in circulating endothelial cells (CEC) and tumor cells (CTC) in patients (pts) receiving bevacizumab and erlotinib for metastatic breast cancer (MBC) predicts stable disease at first evaluation [abstract 525]. J Clin Oncol 2005;23:10s
- [Result] Schippinger W, Lileg B, Ploner F, Weitzer W, Bauernhofer TH, Samonigg H. Neoadjuvant chemotherapy with non-pegylated liposomal doxorubicin, docetaxel and trastuzumab in HER-2/neu overexpressing breast cancer. Ann Oncol 2007; 18 (Suppl 9): 28p
- [Result] Shweiki D, Itin A, Soffer D et al. Vascular endothelial growth factor induced by hypoxia may mediate hypoxia-initiated angiogenesis. Nature (Lond.) 1992; 359: 843-845.Slamon DJ, Clark GM, Wong SG et al. Human breast cancer: correlation of relapse and survival with amplification of the Her-2/neu oncogene. Science 1987; 235:177-182
- [Result] Slamon DJ, Godolphin W, Jones LA, Holt JA, Wong SG, Keith DE, Levin WJ, Stuart SG, Udove J, Ullrich A, et al. Studies of the HER-2/neu proto-oncogene in human breast and ovarian cancer. Science. 1989 May 12;244(4905):707-12. doi: 10.1126/science.2470152.
- [Result] Sledge GW, Miller KD, Moisa CF et al. Safety and efficacy of capecitabine plus bevacizumab as first-line treatment in metastatic breast cancer J Clin Oncol 2007; 25: 35s ASCO abstract 1013
- [Result] Traina TA, Dickler MN, Caravelli JF et al. A phase II trial of letrozole in combination with bevacizumab, an anti-VEGF antibody, in patients with hormone receptor-positive metastatic breast cancer [abstract 2030]. Breast Cancer Res Treat 2005;94:S93
- [Result] Tycznski JE, Bray F and. Parkin DM. Breast cancer in Europe. International Agency for Research on Cancer: European Network of Cancer Registries Cancer Fact Sheet 2002; 2
- [Result] Venturini M, Bighin C, Puglisi F, Olmeo N, Aitini E, Colucci G, Garrone O, Paccagnella A, Marini G, Crino L, Mansutti M, Baconnet B, Barbato A, Del Mastro L. A multicentre Phase II study of non-pegylated liposomal doxorubicin in combination with trastuzumab and docetaxel as first-line therapy in metastatic breast cancer. Breast. 2010 Oct;19(5):333-8. doi: 10.1016/j.breast.2010.01.018. Epub 2010 Feb 24. PMID 20185313
- [Result] Von Minckwitz G, Zielinski C, Maarteense E et al. Capecitabine vs. capecitabine + trastuzumab in patients with HER2-positive metastatic breast cancer progressing during trastuzumab treatment: The TBP phase III study (GBG 26/BIG 3-05). J Clin Oncol 26: 2008 (May 20 suppl; abstr 1025)
- [Result] Yardley DA, Hart L, Badarinath S et al. Preliminary results of a multicenter study of bevacizumab with 3 docetaxel-based adjuvant breast cancer regimens. San Antonio Breast Cancer Symposium, 2007, Poster Presentation
- See also: ABCSG official website — http://www.abcsg.at